CLINICAL TRIAL: NCT04409977
Title: Circadian Changes of the Hypothalamic Activity in Patients Suffering From Cluster Headache
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02389
Record Dates: First submitted 2019-06-26; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Cluster Headache
Keywords: Primary Headache; Trigeminal autonomic cephalgia; functional connectivity
MeSH Terms: conditions — Cluster Headache; Trigeminal Autonomic Cephalalgias

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Patients suffering from cluster headache will be included in this group. When analysing the data, the investigators will distinguish those in the in-bout period from those in the out-bout period. People in this group may participate twice: once in the in-bout and once in the out-bout period.
  Interventions: Diagnostic Test: MRI examination
- Control group: Participants not suffering from cluster headache will be included in this group.
  Interventions: Diagnostic Test: MRI examination

INTERVENTIONS:
Diagnostic Test: MRI examination — Patient will be scanned in the MRI twice, once at noon (+/- 1 hour), once at 1 a.m. (+/- 1 hour). The investigators will search for any changes in functional connectivity, particular regarding the connection between the hypothalamus and pain-processing networks.
  Other Names: quantitative sensory testing (QST)

SUMMARY:
Cluster headache attacks do not occur randomly throughout the day, but have a clear circadian rhythmicity. The aim of this study is to investigate circadian changes of the brain, the autonomic nervous system and pain processing systems.

DETAILED DESCRIPTION:
Cluster headache attacks do not occur randomly throughout the day, but have a clear circadian rhythmicity. The aim of this study is to investigate circadian changes in the functional connectivity, spectroscopy, iron deposition and perfusion of the brain. In addition, we plan to investigate circadian changes in the pain threshold of the brain using quantitative sensory testing (QST). Finally, we will investigate changes in the autonomic nervous system measuring the pupillary response.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cluster headache (CH) may enter the patient group, patients not suffering from CH may enter the control group.
* knowledge of the german language suffices to understand the information sheet and consent form
* having read, understood and signed the consent form

Exclusion Criteria:

* Pregnancy
* contraindications for the MRI scan (particularly metal splinters, ferromagnetic devices and implants)
* claustrophobia
* obesity (MRI > 35 kg/m2)
* shift working (last night shift must date back more than one week)
* jet lag (last travel over more than two time zones must date back more than one week)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from cluster headache.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Circadian rhythmicity of the functional connectivity of the brain | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline in functional connectivity of the brain using whole-brain fMRI

SECONDARY OUTCOMES:
Circadian rhythmicity of the pain threshold | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline of the pain threshold in the face using quantitative sensory testing (QST)
Circadian changes in the perfusion of the brain. | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline in perfusion of the brain using Arterial Spin Labeled MRI Perfusion Imaging and vascular space occupancy sequences
Circadian rhythmicity of the autonomic system | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline in the pupillary response (measured using pupillometry)
Circadian rhythmicity of the spectroscopy of the hypothalamus | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline in the spectroscopy of the hypothalamus
Circadian rhythmicity of the spectroscopy of the hypothalamus | Measurements will be made at noon and at 1 a.m. (+/- 2 hours); we will compare these measurements to identify changes.
  Changes from baseline in the iron concentration of the brain using quantitative susceptibility mapping

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Pohl, MD, Principal Investigator — University of Zurich
Locations (1):
- University hospital Zurich, Zurich, Canton of Zurich, Switzerland